CLINICAL TRIAL: NCT04627922
Title: N-Acetylcysteine for Smoking Cessation in Tobacco and Cannabis Co-Use: A Randomized Controlled Trial
Brief Title: N-Acetylcysteine for Smoking Cessation in Tobacco and Cannabis Co-Use
Acronym: NAC_CUD-TUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ellen Herbst (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor-Investigator, Ellen Herbst, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-31475
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Use; Tobacco Use Disorder; Drug Use Disorder
Keywords: Tobacco; Cannabis; N-acetylcysteine; NAC
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders; Marijuana Abuse | interventions — Acetylcysteine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetyl cysteine (NAC) & cognitive behavioral therapy (Experimental): N-acetyl cysteine (NAC) & cognitive behavioral therapy experimental arm consists of 30 regular cigarette smokers and cannabis users with current TUD, who will be randomized to receive N-acetyl cysteine 3600 mg per day over 8 weeks to experimental arm. Participants will also receive weekly cognitive behavioral therapy for substance use disorders targeting TUD and cannabis use.
  Interventions: Drug: N-Acetyl cysteine; Behavioral: Cognitive behavioral therapy (CBT)
- Placebo Comparator: Placebo & cognitive behavioral therapy (Placebo Comparator): Placebo comparator & cognitive behavioral therapy arm consists of 30 regular cigarette smokers and cannabis users with current TUD, who will be randomized to receive placebo over 8 weeks. Participants will also receive weekly cognitive behavioral therapy for substance use disorders targeting TUD and cannabis use.
  Interventions: Other: Placebo comparator; Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: N-Acetyl cysteine — The investigators will examine N-acetyl cysteine to treat concurrent tobacco use disorder and cannabis use in a double-blind, placebo-controlled RCT. Sixty regular cigarette smokers with current tobacco use disorder and cannabis use will be randomized to receive NAC 3600 mg per day over 8 weeks.
  Other Names: NAC
  Arms: N-acetyl cysteine (NAC) & cognitive behavioral therapy
Other: Placebo comparator — The investigators will examine N-acetyl cysteine to treat concurrent tobacco use disorder and cannabis use in a double-blind, placebo-controlled RCT. Sixty regular cigarette smokers and cannabis users with current tobacco use disorder will be randomized to receive placebo per day over 8 weeks.
  Arms: Placebo Comparator: Placebo & cognitive behavioral therapy
Behavioral: Cognitive behavioral therapy (CBT) — Participants in both groups will receive 8 weekly cognitive behavioral therapy sessions for substance use disorder targeting both tobacco and cannabis use.
  Other Names: CBT

SUMMARY:
Tobacco and cannabis co-use is a common and growing public health problem, especially in states that have legalized cannabis. There are no pharmacologic treatments for co-occurring tobacco and cannabis use. Co-use may make quitting either substance more difficult, given the synergistic effects of cannabis and nicotine on neurobiological systems that mediate reward and shared cues reinforcing co-use. N-acetylcysteine (NAC), an FDA-approved medication and over-the-counter supplement, has shown promise in animal studies and randomized controlled trials (RCTs) in reducing tobacco and cannabis craving and use.

DETAILED DESCRIPTION:
N-acetylcysteine (NAC), an FDA-approved medication and over-the-counter supplement, has shown promise in animal studies and randomized controlled trials (RCTs) in reducing tobacco and cannabis craving and use. NAC's efficacy in treating addiction may be attributable to its central nervous system effects in reducing excessive glutamatergic activity, oxidative stress, and inflammation. NAC has been shown to improve cognition and reduce impulsivity, which in turn may strengthen inhibitory control when presented with contextual cues. To date, no RCT has examined NAC for smoking cessation in the setting of tobacco-cannabis co-use. In a double-blind, placebo-controlled RCT, the investigators will examine a novel pharmacological treatment, NAC, for concurrent tobacco use disorder (TUD) and cannabis use in dual users of tobacco and cannabis. Sixty adult regular cigarette smokers who 1) have smoked 2 cigarettes per day in 15 of the past 30 days, or an average of 1 cigarettes per day for the past 30 days and 2) use cannabis regularly and 3) consent to receive interventions to stop smoking cigarettes and using cannabis will be randomized to receive NAC 3600 mg per day or placebo over 8 weeks. Participants in both groups will receive 8 weekly cognitive behavioral therapy sessions addressing both tobacco and cannabis use. Outcomes will be assessed at Weeks 0, 4, 8, and 12. Primary aims are to determine NAC's efficacy in decreasing cigarette use, nicotine dependence levels, and craving; and cannabis use, and craving. Exploratory aims include examination of changes in neurocognition with NAC and their potential mediational effects on cigarette and cannabis use outcomes.

NAC SUB-STUDY:

Because of the significant clinical and economic burden imposed by tobacco and cannabis use, it is important to understand the mechanism underlying the progression of tobacco (TUD) and cannabis use disorders (CUD) and any potential treatments. TUD and CUD are associated with elevated oxidative stress and chronic inflammation. It has been suggested that patients dependent on these substances have dysregulated markers of oxidation and inflammation, including gluthathione, erythrocyte sedimentation rate (ESR), C-Reactive protein (CRP), Interleukin-6 (IL-6).

In this sub-study, baseline levels of commonly utilized serum markers of oxidation status and inflammation will be measured in 20 adults recruited under the main study, with the option of being a part of the sub-study who also demonstrate concurrent TUD and cannabis use. The correlation will be determined between changes in serum markers of oxidative stress and magnitude of use of cigarettes and cannabis. If successful, the investigator will establish regulatory patterns of oxidative stress and inflammation in TUD and with concurrent cannabis use for the first time, and will implicate oxidative stress and inflammation as playing key roles in the progression and severity of co-occurring TUD and CUD.

ELIGIBILITY:
Inclusion Criteria:

Participants will be male and female smokers ages 18 and over who: 1) have smoked 2 cigarettes per day in 15 of the past 30 days, or an average of 1 cigarettes per day for the past 30 days; 2) endorse the use of cannabis within the past 30 days, reported by TLFB, and have positive urine THC at Week 0 or up to 30 days prior; 3) meet criteria for TUD in the past 12 months per DSM-5, assessed by medical record review and clinical assessment; and 4) consent to receive interventions to stop smoking cigarettes and reducing cannabis use. Although co-users can use tobacco and cannabis simultaneously (i.e. in "spliffs") and other forms of nicotine and tobacco, participants must smoke combustible cigarettes that are not mixed with cannabis on a daily basis to participate. Individuals of childbearing potential (ages 18-55) must have a negative urine pregnancy test at the time of screening. Individuals who have been prescribed bupropion for depression, not smoking cessation, are eligible to participate in this study. All participants must be California residents (Veterans enrolled in VA healthcare in another state are eligible).

Exclusion Criteria:

1) Psychotic disorders, bipolar disorder, neurocognitive disorder, or other psychiatric or medical conditions judged by the PI to be unstable in the past 30 days, based on screening results and/or medical record review. 2) Concurrent participation in another pharmacological tobacco cessation study. 3) Individuals who are pregnant or lactating. 4) Non-study NAC use at enrollment or at any time during the study period. 5) Use of medications for TUD (NRT, bupropion, or varenicline) at enrollment or at any time during the study period. 6) A suicide attempt or suicidal ideation with intent in the 30 days prior to enrollment. 7) Non-residents of California or Veterans in another state who are not enrolled in VA healthcare.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with reported drug usage | Baseline
  Participants will participate in urine drug testing which may screen for multiple substances, including amphetamines, methamphetamine, benzodiazepines, barbiturates, marijuana, cocaine, opiates, Phencyclidine (PCP), methadone, nicotine, and alcohol throughout the course of the study. An encrypted email will be sent from VA-protected email accounts from study staff to request an encrypted response with an attached photo image of results. There will be clear instructions to encrypt a de-identified image results message, and the collection of identifying information will not be allowed.
Number of participants with reported drug usage | 4 weeks
  Participants will participate in urine drug testing which may screen for multiple substances, including amphetamines, methamphetamine, benzodiazepines, barbiturates, marijuana, cocaine, opiates, Phencyclidine (PCP), methadone, nicotine, and alcohol throughout the course of the study. An encrypted email will be sent from VA-protected email accounts from study staff to request an encrypted response with an attached photo image of results. There will be clear instructions to encrypt a de-identified image results message, and the collection of identifying information will not be allowed.
Number of participants with reported drug usage | 8 weeks
  Participants will participate in urine drug testing which may screen for multiple substances, including amphetamines, methamphetamine, benzodiazepines, barbiturates, marijuana, cocaine, opiates, Phencyclidine (PCP), methadone, nicotine, and alcohol throughout the course of the study. An encrypted email will be sent from VA-protected email accounts from study staff to request an encrypted response with an attached photo image of results. There will be clear instructions to encrypt a de-identified image results message, and the collection of identifying information will not be allowed.
Number of participants with reported drug usage | 12 weeks
  Participants will participate in urine drug testing which may screen for multiple substances, including amphetamines, methamphetamine, benzodiazepines, barbiturates, marijuana, cocaine, opiates, Phencyclidine (PCP), methadone, nicotine, and alcohol throughout the course of the study. An encrypted email will be sent from VA-protected email accounts from study staff to request an encrypted response with an attached photo image of results. There will be clear instructions to encrypt a de-identified image results message, and the collection of identifying information will not be allowed.
Mean Salivary Cotinine Levels | 4 weeks
  For participants who report not smoking, a saliva sample will be collected to determine salivary cotinine levels at each visit. Cotinine levels are an established method to biochemically verify a participants smoking status.
Mean Salivary Cotinine Levels | 8 weeks
  For participants who report not smoking, a saliva sample will be collected to determine salivary cotinine levels at each visit. Cotinine levels are an established method to biochemically verify a participants smoking status.
Mean Salivary Cotinine Levels | 12 weeks
  For participants who report not smoking, a saliva sample will be collected to determine salivary cotinine levels at each visit. Cotinine levels are an established method to biochemically verify a participants smoking status.
Change in Percentage of Participants with Point Prevalent Abstinence | Up to 12 weeks
  Seven-day point prevalence cigarette abstinence will be defined as the percentage of participants who have reported no smoking or nicotine use on the 7 consecutive days prior to the assessment with biochemically verified cotinine levels of < 10 nanograms/ milliliter.
Changes in Score on the Contemplation Ladder | Up to 12 weeks
  The Contemplation Ladder is a visual analog comprised of 11 rungs and 5 anchor statements, representing stages of change. The response options (0) to (3) corresponded with the stage of precontemplation, (4) to (6) represented the stage of contemplation, (7) and (8) referred to the stage of preparation, (9) and (10) represented the stage of action and stage of maintenance respectively. It is a brief measure of motivation or readiness to change, where (0) is the least motivated and (10) is the most motivated. This measure has been validated for cigarette and other substance use. This measure will be administered twice at each time point both before and after an activity to assess motivation to stop 1) cigarettes and 2) cannabis.
Change in Scores on the Fagerstrom Test for Nicotine Dependence (FTND) | Up to 12 weeks
  The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Change in Scores on the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) | Up to 12 weeks
  The MTWS-R features two separate measures for examining the severity of nicotine withdrawal symptoms in a participant: a self-report scale and an observer scale. The observer scale asks the scale-taker to rate the severity of four symptoms in someone the they know who is experiencing nicotine withdrawal: "angry/irritable/frustrated," "anxious/tense," "depressed," and "restless/impatient." The self-report version asks for rankings of the severity of those same four symptoms, plus eleven others that cannot be observed by outsiders (including such things as "desire or craving to smoke," "insomnia, sleep problems, awakening at night," or "dizziness). Both scales use a Likert-type scale for the severity ratings, ranging from 0 ("not at all") to 4 ("severe"). These scores are tallied to calculate an a total withdrawal discomfort score.
Change in Scores on the Questionnaire on Smoking Urges (QSU-Brief): Desire to smoke | Up to 12 weeks
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and scores are calculated by summing the item scores
Change in Scores on the Questionnaire on Smoking Urges (QSU-Brief): Nicotine withdrawal | Up to 12 weeks
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and scores are calculated by summing the item scores
Change in Scores on the Questionnaire on Smoking Urges (QSU-Brief): Total | Up to 12 weeks
  The QSU-Brief consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and total scores are calculated by summing the item scores.
Change in Scores on the Cannabis Use Disorder Identification Test - Revised (CUDIT-R) | Up to 12 weeks
  This questionnaire was designed for self-administration and is scored by adding each of the 8 items relating to cannabis use over the past six months. Question 1-7 are scored on a 0-4 scale Question 8 is scored 0,2, or 4. Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
Change in Scores on the Marijuana Craving Questionnaire Short Form (MCQ-SF) Total | Up to 12 weeks
  This 12-item multidimensional measure assesses cannabis craving based on 4 factors: Compulsivity, Emotionality, Expectancy, Purposefulness. Each item asks about the respondent's feelings and thoughts about smoking marijuana as he or she is completing the questionnaire (i.e., right now). Each response is scored a number ranging from 1 (strongly disagree) to 7 (strongly agree) and scores are using the mean to the corresponding item. Total Scores are the sum of the means for the 4 subscales.
Change in Scores on the Cannabis Withdrawal Scale | Up to 12 weeks
  This questionnaire is a copyrighted, validated, 19-item assessment of cannabis withdrawal symptoms. Higher total Score is indicative of increasing or decreasing severity of withdrawal
Change in Scores on the Beck Depression Inventory (BDI) | Up to 12 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Each question had a set of at least four possible responses When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows: 0-9 minimal depression, 10-18 indicates mild depression, 19-29 indicates moderate depression, 30-63 indicates severe depression. Higher total scores indicate more severe depressive symptoms.
Change in Scores on the Beck Anxiety Inventory (BAI) | Up to 12 weeks
  The BAI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of anxiety. Each question had a set of at least four possible responses When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the anxiety severity. The standard cut-off scores were as follows: 0-9 minimal anxiety, 10-18 indicates mild anxiety, 19-29 indicates moderate anxiety, 30-63 indicates severe anxiety. Higher total scores indicate more severe anxiety symptoms.
Change in Scores on the Emotion Regulation Questionnaire (ERQ) | Up to 12 weeks
  The ERQ is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Items 1, 3, 5, 7, 8, 10 make up the Cognitive Reappraisal facet.
  Items 2, 4, 6, 9 make up the Expressive Suppression facet and scores can be summed to create a total score. Higher scores indicate a greater ability for participants to regulate their emotions.
Change in Scores on the Mindful Attention Awareness Scale (MAAS) | Up to 12 weeks
  The MAAS is a 15-item scale measuring dispositional mindfulness by asking respondents' to indicate how frequently they experience mindlessness (i.e., "I run through activities without being really attentive to them") on a 6-point Likert-type scale ranging from 1 (almost always) to 6 (almost never). To score the MAAS, a mean of the 15 items is calculated. Higher scores reflect higher levels of dispositional mindfulness. With these higher scores also come lower reported negative emotional states.
Change in Scores on the Client Satisfaction Questionnaire (CSQ-8) | Up to 12 weeks
  The CSQ-8 is an 8 item measure that will be utilized to measure the satisfaction with the manualized treatment. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — San Francisco Veterans Affairs Medical Center; Madeline Martinez Rivas, PhD, Study Director — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schauer GL, Berg CJ, Kegler MC, Donovan DM, Windle M. Assessing the overlap between tobacco and marijuana: Trends in patterns of co-use of tobacco and marijuana in adults from 2003-2012. Addict Behav. 2015 Oct;49:26-32. doi: 10.1016/j.addbeh.2015.05.012. Epub 2015 May 23. PMID 26036666
- [Background] Davis CN, Slutske WS, Martin NG, Agrawal A, Lynskey MT. Identifying subtypes of cannabis users based on simultaneous polysubstance use. Drug Alcohol Depend. 2019 Dec 1;205:107696. doi: 10.1016/j.drugalcdep.2019.107696. Epub 2019 Oct 28. PMID 31726429
- [Background] Eisenlohr-Moul TA, Peters JR, Pond RS Jr, DeWall CN. Both trait and state mindfulness predict lower aggressiveness via anger rumination: A multilevel mediation analysis. Mindfulness (N Y). 2016 Jun;7(3):713-726. doi: 10.1007/s12671-016-0508-x. Epub 2016 Mar 9. PMID 27429667
- [Derived] Herbst ED, Pennington DL, Borsari B, Manuel J, Yalch M, Alcid E, Martinez Rivas M, Delacruz J, Rossi N, Garcia B, Wong N, Batki SL. N-acetylcysteine for smoking cessation among dual users of tobacco and cannabis: Protocol and rationale for a randomized controlled trial. Contemp Clin Trials. 2023 Aug;131:107250. doi: 10.1016/j.cct.2023.107250. Epub 2023 Jun 2. PMID 37271412
- See also: Provides Link to NAC Study (in development) — https://addictionresearch.ucsf.edu/